CLINICAL TRIAL: NCT00259792
Title: A Comparison of Symbicort Single Inhaler and Conventional Best Practice for the Treatment of Persistent Asthma in Adolescents and Adults - a 26-week, Randomised, Open, Parallel Group Multicentre Study
Brief Title: SYMPHONIE - A Comparison of Symbicort Single Inhaler and Conventional Best Practice for the Treatment of Persistent Asthma in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00005; SYMPHONIE
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol Turbuhaler
  Other Names: Symbicort

SUMMARY:
The purpose of the study is to compare the efficacy of a flexible dose of Symbicort with conventional stepwise treatment according to asthma treatment guidelines in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 3 months history of asthma, diagnosed according to the American Thoracic Society (ATS) definition. Prescribed inhaled GCS at a dose of ³400 µg/day and within the approved label for the relevant drug during the last 3 months prior to Visit 1.

Exclusion Criteria:

* Use of any b-blocking agent, including eye-drops, Use of oral GCS as maintenance treatment, A history of smoking ³ 10 pack years (1 pack year = 1 pack (20 cigarettes) per day for one year or equivalent).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of asthma exacerbations, Mean use of as-needed medication, Prescribed asthma medication, Asthma Control Questionnaire, Satisfaction with Asthma Treatment Questionnaire, Safety: Serious Adverse Events and discontinuations due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (82):
- France (82):
  - Research Site, Abbeville
  - Research Site, Agen
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alès
  - Research Site, Ambérieu-en-Bugey
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Apt
  - Research Site, Arles
  - Research Site, Aubagne
  - Research site, Avignon
  - Research Site, Avrillé
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Blois
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourgoin
  - Research Site, Brest
  - Research Site, Briey
  - Research Site, Bron
  - Research Site, Cabestany
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cambrai
  - Research Site, Carcassonne
  - Research Site, Castelnau-le-Lez
  - Research site, Challans
  - Research Site, Champs-sur-Marne
  - Research Site, Charleville-Mézières
  - Research Site, Châlons-en-Champagne
  - Research Site, Chelles
  - Research Site, Cherbourg Octeville
  - Research Site, Chevilly-Larue
  - Research Site, Choisy-le-Roi
  - Research site, Cholet
  - Research Site, Colmar
  - Research Site, Cornebarrieu
  - Research Site, Courbevoie
  - Research Sites, Créteil
  - Research Site, Denain
  - Research Site, Dieppe
  - Research Site, Dijon
  - Research Site, Dole
  - Research Site, Ermont
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Étampes
  - Research Site, Fécamp
  - Research Site, Forbach
  - Research Site, Gournay-sur-Marne
  - Research Site, Grenoble
  - Research Site, Hagondange
  - Research Site, Hazebrouck
  - Research Site, Herblay-sur-Seine
  - Research Site, Hénin-Beaumont
  - Research Site, Hyères
  - Research Site, Issy-les-Moulineaux
  - Research Site, Joigny
  - Research Site, Juan-les-Pins
  - Research Site, La Roche-sur-Yon
  - Research site, La Rochelle
  - Research Site, La Teste-de-Buch
  - Research Site, Lagardelle-sur-Lèze
  - Research Site, Le Havre
  - Research Site, Le Puy-en-Velay
  - Research site, Lens
  - Research Site, Les Mureaux
  - Research Site, Libourne
  - Research Site, Lille
  - Research site, Limoges
  - Research site, Loudéac
  - Research site, Lunéville
  - Research Site, Lyon
  - Research Site, Marcq-en-Barœul